CLINICAL TRIAL: NCT02686710
Title: Comparison of the Effects of TIVA vs VIMA on Content of GSK-3beta in Leucocytes in On-pump Patients: a Randomized Clinical Trial
Brief Title: Comparison of the Effects of TIVA vs VIMA on Content of GSK-3beta in Leucocytes in On-pump Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Moscow Regional Research and Clinical Institute (MONIKI) (Other Government)
Responsible Party: Principal Investigator, Valery V. Likhvantsev, Professor, senior researcher, Moscow Regional Research and Clinical Institute Moniki n.a. M.F. Vladimirskiy, Moscow Regional Research and Clinical Institute (MONIKI)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GSK-TV-L
Record Dates: First submitted 2016-02-16; First posted 2016-02-19 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Glycogen Synthase Kinase 3
MeSH Terms: interventions — Sevoflurane; Propofol

ARMS (3):
- VIMA (Active Comparator): Patiens receiving volatile induction and maitenance of anesthesia
  Interventions: Drug: Sevoflurane
- TIVA (Active Comparator): Patiens receiving total intravenous anesthesia based on propofol
  Interventions: Drug: Propofol
- Combi (Active Comparator): Patiens receiving total intravenous induction and volatile anesthesia
  Interventions: Drug: Sevoflurane; Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane
  Arms: Combi; VIMA
Drug: Propofol
  Arms: Combi; TIVA

SUMMARY:
Assessment of GSK-3beta contents in leukocytes in on-pump cardiosurgical patients receiving either volatile or intravenous anesthesia

ELIGIBILITY:
Inclusion Criteria:

elective on-pump CABG

Exclusion Criteria:

re-operation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Gsk-3beta base line content | base line
Gsk-3beta content after induction | 20 minutes after tracheal intubation
Gsk-3beta content after surgery | immediately after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Moscow Regional Research and Clinical Institute Moniki n.a. M.F. Vladimirskiy, Moscow, Russia